CLINICAL TRIAL: NCT06664762
Title: Left Lateral Position Versus Supine Position in Colonoscopy, a Multicenter Single-blind Randomized Clinical Trial Study
Brief Title: Left Lateral Position Versus Supine Position in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Collaborators: Hospital Civil Juan I. Menchaca (Other); Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Roberto Ulises Cruz Neri, Principal investigator, Master in Science, Medical Staff in Coloproctology Department at Hospital Civil Fray Antonio Alcalde, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 150/24
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: multicenter single-blind randomized clinical trial study
Who Masked: Care Provider
Masking Description: The main investigators will be in charge of randomizing all the patients ellegible for this protocol, and the care providers and endoscopists will be masked when it comes to knowing to which arm of the study each patient belongs to, untill the moment they need to perform the colonoscopy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left lateral position during colonoscopy (Active Comparator)
  Interventions: Behavioral: Left lateral position intervention
- Supine position during colonoscopy (Active Comparator)
  Interventions: Behavioral: Supine position intervention

INTERVENTIONS:
Behavioral: Left lateral position intervention — Patients will be randomized and asigned to start and remain in left lateral position during the colonoscopy
  Arms: Left lateral position during colonoscopy
Behavioral: Supine position intervention — Patients will be randomized and asigned to start and remain in supine position during the colonoscopy
  Arms: Supine position during colonoscopy

SUMMARY:
Currently, colonoscopy is a minimally invasive method that can be used as a diagnostic and therapeutic method by endoscopists, gastroenterologists and coloproctologists. Due to the importance and big impact this method has, it is necessary to both optimize its efficiency, and improve its quality, which is one of the main objectives of this protocol.

By observing which position its faster and which one also results in fewer complications when performing a colonoscopy without reducing its performance and following all the internationally established quality standards regarding colonoscoscopy.

The risk of this protocol implies a risk no greater than the minumum the procedure itself has, and does not generate extra cost for all of the patients subjected to this protocol.

DETAILED DESCRIPTION:
Currently, colonoscopy is one of the most used procedures when it comes to the study and treatment of patients with gastrointestinal conditions, including colorectal cancer, inflammatory bowel disease, etc.

In the area of colorectal neoplasia, colonoscopy has three main functions, which are to diagnose the desease itself and prevent its development by detecting and eliminating potentially premalignant lesions, as well as providing a diagnosis of cancer at an early stage.

The effectiveness of colonoscopy is crucial to carry out an accurate examination of the entire colorectal mucosa, which is why the quality of the procedure has been a subject of study in recent years. Among multiple factors that influence the quality of colonoscopies, the investigators can mention intestinal preparation, which is essential for an accurate procedure, because if patients have an inadequate preparation, it could impair the detection of lesions, since usually, in patients with little or no preparation, colonoscopy can be either incomplete, which requires the study to be repeated, or in case the study continues despite poor intestinal preparation, the presence of feces implies poor visualization of the colonic mucosa, which reduces the ability to detect lesions such as polyps, especially if they are <5 mm. Therefore, the type of solution and tolerability, the preparation regimen and the moment in which the intestinal preparation is performed are considerations to evaluate when performing a colonoscopy.

The position during the colonoscopy is another factor that can influence colonoscopy´s effectiveness, and also, the main focus for the investigators to study. Traditionally, if no position changes occur during colonoscopy, it begins and ends in the left lateral position. However, recent evidence suggests that supine position may reduce the disadvantages of the left lateral position, through decreased frequency of position changes and decreased abdominal pressure, which may result in an easier endoscope insertion in supine position when comparing it to left lateral position, however, there is very few information on the optimal insertion technique in colonoscopy, but it has been observed that in left lateral position, the air leaves the left colon causing it to collapse and also creating sharp curves that can be difficult to overcome during the procedure.

As previously mentioned, colonoscopy insertion is technically challenging, and one of the few clinical trials available that targeted the determination of optimal patient positioning during colonoscopy insertion compared the supine starting position with the left lateral starting position, and the investigators found that cecal intubation times decreased and patient comfort scores improved when using the supine position.

Therefore, patient positioning in colonoscopy has been proposed as a simple and inexpensive technique to increase luminal distension and improve navigation through the colon. Based on what has been mentioned before, using the initial supine position could be a convenient method to reduce cecal intubation time, reduce pain, and improve acceptance of colonoscopy among patients. However, more research is necessary in this area to stablish the advantages of the initial supine position over other positions thar are classically used.

Based on everything that has been described above, the investigators asked themselves the following research question to start this clinical trial: Is there a significant difference in the effectiveness and comfort of performing colonoscopy, when comparing the left lateral position with the supine position?

The institutes where this clinical trial will take place have subjects for study that are ellegible to enroll as participants, infraestructure and health care providers trained to perform colonoscopies and a complete investigators team to collect and analyze the data for this protocol.

The protocol will be limited only to patients who are beneficiaries of each of the hospitals involved. Furthermore, as it is a single-blind randomized clinical trial, the endoscopists in the study cannot be blinded, so investigator bias will not be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for colonoscopy in our coloproctology service
* Both women and men
* Patients within an age range of 18-79 years
* Patients who agree having a colonoscopy and who sign the informed consent to participate in the protocol

Exclusion Criteria:

* Patients under 18 or over 80 years old
* All patients that won´t like to participate in the protocol or won´t sign the informed consent
* Pregnant women
* Patients with a medical record of colonic resection, ostomy status, severe cardiopulmonary and renal diseases, major psychiatric disorders, therapeutic colonoscopy or any contraindications for colonoscopy
* Non compliance with the colonic preparation regimen
* Active bleeding during the procedure
* Patients with a known diagnosis of colorectal cancer
* Patients with class III obesity

Elimination criteria:

* Boston score <6 for colonic preparation
* Patients with a colonic lesion that makes it difficult to pass the colonoscope
* Patients with insufficient sedation that requires the procedure to stop temporarily
* Bowel perforation during colonoscopy
* Inability to reach the cecum despite loop reduction maneuvers
* Indication to suspend the study given by the anesthesiologist

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Arrival time to the cecum | From date of randomization until the colonoscopy is done, assessed up to 9 months
ileocecal valve intubation time | From date of randomization until the colonoscopy is done, assessed up to 9 months

SECONDARY OUTCOMES:
Percentage of ileocecal valve intubation | From date of randomization until the colonoscopy is done, assessed up to 9 months
Adenoma detection rate | From date of randomization until the colonoscopy is done, assessed up to 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- Mexico (3):
  - Antigüo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Nuevo Hospital Civil de Guadalajara "Juan I. Menchaca", Guadalajara, Jalisco
  - IMSS Hospital General Regional 220 "José Vicente Villada", México, Toluca de Lerdo

REFERENCES:
- [Background] de la Torre Bravo A. [The astonishing evolution of endoscopy]. Rev Gastroenterol Mex. 2001 Jan-Mar;66(1):58-9. No abstract available. Spanish. PMID 11464632
- [Background] Spaner SJ, Warnock GL. A brief history of endoscopy, laparoscopy, and laparoscopic surgery. J Laparoendosc Adv Surg Tech A. 1997 Dec;7(6):369-73. doi: 10.1089/lap.1997.7.369. PMID 9449087
- [Background] Antoniou SA, Antoniou GA, Koutras C, Antoniou AI. Endoscopy and laparoscopy: a historical aspect of medical terminology. Surg Endosc. 2012 Dec;26(12):3650-4. doi: 10.1007/s00464-012-2389-y. Epub 2012 Jun 21. PMID 22717798
- [Background] Irving MH, Catchpole B. ABC of colorectal diseases. Anatomy and physiology of the colon, rectum, and anus. BMJ. 1992 Apr 25;304(6834):1106-8. doi: 10.1136/bmj.304.6834.1106. No abstract available. PMID 1586826
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Neilson LJ, Bevan R, Panter S, Thomas-Gibson S, Rees CJ. Terminal ileal intubation and biopsy in routine colonoscopy practice. Expert Rev Gastroenterol Hepatol. 2015 May;9(5):567-74. doi: 10.1586/17474124.2015.1001744. Epub 2015 Jan 12. PMID 25582839
- [Background] Vergis N, McGrath AK, Stoddart CH, Hoare JM. Right Or Left in COLonoscopy (ROLCOL)? A Randomized Controlled Trial of Right- versus Left-Sided Starting Position in Colonoscopy. Am J Gastroenterol. 2015 Nov;110(11):1576-81. doi: 10.1038/ajg.2015.298. Epub 2015 Sep 29. PMID 26416195
- [Background] Vergis N, Scarborough AJ, Morris JA, Hoare JM. Prone or Left for Colonoscopy? A Randomized Controlled Trial of Prone Versus Left-sided Starting Position for Colonoscopy. J Clin Gastroenterol. 2018 Nov/Dec;52(10):e82-e86. doi: 10.1097/MCG.0000000000000871. PMID 28644314
- [Background] Zhao S, Yang X, Meng Q, Wang S, Fang J, Qian W, Xia T, Pan P, Wang Z, Gu L, Chang X, Zou D, Li Z, Bai Y. Impact of the supine position versus left horizontal position on colonoscopy insertion: a 2-center, randomized controlled trial. Gastrointest Endosc. 2019 Jun;89(6):1193-1201.e1. doi: 10.1016/j.gie.2019.01.009. Epub 2019 Jan 18. PMID 30660634
- [Background] Chokshi RV, Hovis CE, Hollander T, Early DS, Wang JS. Prevalence of missed adenomas in patients with inadequate bowel preparation on screening colonoscopy. Gastrointest Endosc. 2012 Jun;75(6):1197-203. doi: 10.1016/j.gie.2012.01.005. Epub 2012 Feb 28. PMID 22381531
- [Background] Cappell MS, Friedel D. The role of sigmoidoscopy and colonoscopy in the diagnosis and management of lower gastrointestinal disorders: technique, indications, and contraindications. Med Clin North Am. 2002 Nov;86(6):1217-52. doi: 10.1016/s0025-7125(02)00076-7. PMID 12510453
- [Background] Gangwani MK, Aziz A, Dahiya DS, Nawras M, Aziz M, Inamdar S. History of colonoscopy and technological advances: a narrative review. Transl Gastroenterol Hepatol. 2023 Apr 20;8:18. doi: 10.21037/tgh-23-4. eCollection 2023. PMID 37197258
- [Background] Church J. Colonoscopy: what are we missing? Surg Oncol Clin N Am. 2014 Jan;23(1):1-9. doi: 10.1016/j.soc.2013.09.001. Epub 2013 Nov 1. PMID 24267161
- [Background] Greene A, Borgoankar M, Hodgkinson K, Garland C, Bacque L, Pace D. A randomized controlled trial comparing right and left lateral decubitus starting position on outcomes in colonoscopy. Surg Endosc. 2020 Aug;34(8):3656-3662. doi: 10.1007/s00464-020-07661-x. Epub 2020 May 26. PMID 32458286